CLINICAL TRIAL: NCT06365853
Title: A Randomized Phase 2 Study of Ocular Toxicity Evaluation and Mitigation During Treatment With Mirvetuximab Soravtansine in Patients With Recurrent Ovarian Cancer With High Folate Receptor-Alpha Expression
Brief Title: A Study of Ocular Toxicity Evaluation and Mitigation During Treatment With Mirvetuximab Soravtansine in Participants With Recurrent Ovarian Cancer With High Folate Receptor-Alpha Expression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0424; 2023-505617-24-00 (Other: EU CT)
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Ovarian Cancer; Folate Receptor-Alpha Positive
MeSH Terms: conditions — Ovarian Neoplasms | interventions — mirvetuximab soravtansine; Lubricant Eye Drops; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary Prophylactic Steroid Eye Drops (Experimental): Prednisolone acetate ophthalmic suspension 1% 6 times daily on Days -1 to 4 and 4 times daily (QID) on Days 5 to 8 of each cycle; Lubricating eye drops QID throughout the entire cycle (doses should follow steroid dosing, when given, by approximately 15 minutes); MIRV 6 milligrams (mg)/kilogram (kg) adjusted ideal body weight (AIBW) every 3 weeks (Q3W) on Day 1 of each cycle. Each cycle length = 21 days.
  Interventions: Drug: Mirvetuximab Soravtansine; Drug: Lubricating Eye Drops; Drug: Prednisolone acetate ophthalmic suspension 1% eye drops
- Primary Prophylactic Vasoconstricting Eye Drops (Experimental): Primary prophylactic brimonidine tartrate ophthalmic solution eye drops 3 times daily (TID) on Days 1 to 8 of each cycle (vasoconstricting drops should be started on the day of first infusion and should begin before the first infusion on Cycle 1 Day 1); Lubricating eye drops QID throughout the entire cycle (doses should follow brimonidine dosing, when given, by approximately 15 minutes); MIRV 6 mg/kg AIBW Q3W on Day 1 of each cycle. Each cycle length = 21 days.
  Interventions: Drug: Mirvetuximab Soravtansine; Drug: Lubricating Eye Drops; Drug: Brimonidine tartrate ophthalmic solution eye drops

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine — Mirvetuximab soravtansine is an antibody drug conjugate designed to target folate receptor α (FRα). It consists of the humanized anti-FRα monoclonal antibody (mAb) M9346A attached via a cleavable disulfide linker to the cytotoxic maytansinoid, DM4.
  Other Names: IMGN853; MIRV
Drug: Lubricating Eye Drops — Lubricating artificial tears should be administered at least 15 minutes after corticosteroid or brimonidine eye drop administration.
Drug: Prednisolone acetate ophthalmic suspension 1% eye drops — Self-administration of prednisolone acetate ophthalmic suspension 1% eye drops as prescribed by the treating physician.
  Arms: Primary Prophylactic Steroid Eye Drops
Drug: Brimonidine tartrate ophthalmic solution eye drops — Self-administration of brimonidine tartrate ophthalmic solution eye drops as prescribed by the treating physician.
  Arms: Primary Prophylactic Vasoconstricting Eye Drops

SUMMARY:
The purpose of this study is to evaluate the incidence rate and severity of prespecified mirvetuximab soravtansine (MIRV)-related ocular treatment-emergent adverse events (TEAEs) and assess prophylaxis strategies in all participants (symptomatic and asymptomatic) undergoing prospective ophthalmic evaluation with recurrent ovarian cancer (participants with either platinum-sensitive ovarian cancer [PSOC] or platinum-resistant ovarian cancer [PROC]) with high folate receptor alpha (FRα) expression.

DETAILED DESCRIPTION:
Participants will be randomized (1:1) to 1 of 2 ocular adverse event (AE) risk mitigation strategy arms (primary prophylactic steroid eye drops versus primary prophylactic vasoconstricting eye drops).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of epithelial ovarian, fallopian tube, and primary peritoneal cancer (EOC) with high FRα expression.
* Participant's tumor must be FRα positive (FRα high) as defined by either the VENTANA FOLR1 (FOLR-2.1) IUO Assay, or the VENTANA FOLR1 ( FOLR1-2.1) RxDx Assay (hereafter collectively termed VENTANA FOLR1 Assay) (≥ 75% cells exhibit ≥ 2+ membrane staining intensity).
* Participants with known breast cancer susceptibility gene (BRCA) mutations (tumor or germline) must have received poly (ADP-ribose) polymerase inhibitors (PARPi).
* Participants must have completed prior therapy within the specified times below:

  1. Systemic antineoplastic therapy ≥ 5 half-lives or 4 weeks (whichever is shorter) before first dose of MIRV;
  2. Focal radiation completed ≥ 2 weeks before the first dose of MIRV.
* Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities (except alopecia).
* Women of childbearing potential (WOCBP) must agree to use highly effective contraceptive method(s) while on MIRV and for ≥ 7 months after the last dose; and must have a negative pregnancy test ≤ 4 days before the first dose of MIRV.

Exclusion Criteria:

* Participants with borderline ovarian tumor or non-epithelial histology or mixed histology including borderline or non-epithelial histology will be excluded.
* PROC participants with primary platinum-refractory disease, defined as disease that did not respond to (complete response [CR] or partial response [PR]) or progressed within ≤ 3 months of the last dose of first line platinum-containing chemotherapy.
* Participants with > Grade 1 peripheral neuropathy per National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0).
* Participants with significant active or chronic corneal disorders (for example, corneal dystrophies, degenerations, limbal stem cell deficiency), history of corneal transplantation, significant ocular inflammatory conditions (for example, active or recurrent uveitis), or other active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, active diabetic retinopathy with macular edema, macular degeneration requiring treatment ≤ 90 days before first dose, presence of papilledema, best corrected visual acuity (BCVA) worse than 20/70 in either eye, or monocular vision.
* Participants receiving corticosteroid or vasoconstricting eyedrops at baseline or within 5 weeks of Cycle 1 Day 1.
* Participants who received prior treatment with MIRV or other FRα-targeting agents. Note: Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With MIRV-related Corneal TEAEs (≥ Grade 2) in Asymptomatic Participants | Cycle 1 Day 1 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
  This endpoint will be assessed in the participants receiving MIRV who are asymptomatic .

SECONDARY OUTCOMES:
Number of Participants With Ocular symptom TEAEs in Participants Using Corticosteroid or Vasoconstricting Eye Drop Primary Prophylaxis | Cycle 1 Day 1 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days
Number of Participants With MIRV-related Corneal TEAEs in Symptomatic Participants | Cycle 1 Day 1 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
Number of Participants With Ocular exam TEAEs in Asymptomatic Participants and Symptomatic participants | Cycle 1 Day 1 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
Number of Participants With MIRV-related Corneal TEAEs (≥ Grade 2) in Participants Using Corticosteroid or Vasoconstricting Eye Drop Primary Prophylaxis | Cycle 1 Day 1 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
Number of Participants with ocular exam TEAEs in Participants using corticosteroid or vasoconstricting eye drop primary prophylaxis | Cycle 1 Day 1 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) Composite Score | At Cycle 5 Day 1 or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
Area Under the Curve (AUC) of MIRV | Day 1 and Day 8 of Cycles 1 through 4 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
Maximum Serum Concentration (Cmax) of MIRV | Day 1 and Day 8 of Cycles 1 through 4 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)
Trough Concentration (Ctrough) of MIRV | Day 1 and Day 8 of Cycles 1 through 4 up to 18 weeks or at the 30-day follow-up visit, whichever is earlier (cycle length = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (40):
- United States (12):
  - University of California Los Angeles /ID# 269339, Los Angeles, California
  - Norton Cancer Institute - St. Matthews /ID# 269070, Louisville, Kentucky
  - Holy Cross Hospital - Silver Spring /ID# 269344, Silver Spring, Maryland
  - Mercy David C. Pratt Cancer Center /ID# 269350, St Louis, Missouri
  - The Center Of Hope /ID# 269348, Reno, Nevada
  - Holy Name Medical Center /ID# 269340, Teaneck, New Jersey
  - New York Oncology Hematology - Albany Cancer Center /ID# 269345, Albany, New York
  - Women'S Cancer Care Associates /ID# 269980, Albany, New York
  - Duke Cancer Institute /ID# 269342, Durham, North Carolina
  - Summa Health /ID# 269349, Akron, Ohio
  - UT Southwestern Medical Center /ID# 269341, Dallas, Texas
  - Memorial Hermann Southeast Hospital /ID# 269347, Houston, Texas
- Australia (3):
  - Blacktown Hospital /ID# 269305, Blacktown, New South Wales
  - Newcastle Private Hosptial /ID# 269306, Lambton Heights, New South Wales
  - Monash Health - Monash Medical Centre /ID# 269304, Clayton, Victoria
- Belgium (6):
  - Universitair Ziekenhuis Antwerpen /ID# 269310, Edegem, Antwerpen
  - OLV Ziekenhuis Aalst /ID# 269311, Aalst, Oost-Vlaanderen
  - AZ Sint-Lucas /ID# 269307, Ghent, Oost-Vlaanderen
  - UZ Gent /ID# 269309, Ghent, Oost-Vlaanderen
  - UZ Leuven /ID# 269308, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 269312, Liège
- Canada (3):
  - Universite de Montreal - Hopital Maisonneuve-Rosemont /ID# 268862, Montreal, Quebec
  - Centre Hospitalier De L'Universite De Montreal - Hopital Saint-Luc /ID# 269314, Montreal, Quebec
  - McGill University Health Centre - Glen Site. /ID# 269313, Montreal, Quebec
- France (6):
  - Institut Paoli-Calmettes /ID# 269648, Marseille, Bouches-du-Rhone
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau /ID# 269301, Tours, Indre-et-Loire
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 269330, Paris, Paris
  - Hospices Civils de Lyon - Centre Hospitalier Lyon-Sud /ID# 269327, Pierre-Bénite, Rhone
  - Clinique Victor Hugo Le Mans /ID# 269985, Le Mans, Sarthe
  - GH Diaconesses Croix Saint-Simon /ID# 269329, Paris
- Ireland (2):
  - Mater Misericordiae University Hospital /ID# 269334, Dublin
  - Beaumont Hospital /ID# 268864, Dublin
- Spain (8):
  - Hospital San Pedro de Alcántara /ID# 269320, Cáceres, Caceres
  - Hospital Universitario de Jaén /ID# 269319, Jaén, Jaen
  - Usp Instituto Universitario Dexeus /ID# 269322, Barcelona
  - Hospital Universitario Vall de Hebron /ID# 269315, Barcelona
  - Hospital Universitario Ramon y Cajal /ID# 269318, Madrid
  - Hospital Universitario 12 de Octubre /ID# 269321, Madrid
  - Hospital Universitario La Paz /ID# 269302, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 269325, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=IMGN853-0424